CLINICAL TRIAL: NCT00044993
Title: Phase II, Single Arm, Single Institution Clinical Trial of Docetaxel and Doxorubicin in Combination With Local Administration of INGN 201 (Ad5CMV-p53) in Locally Advanced Breast Cancer (LABC)
Brief Title: Chemotherapy Combined With Gene Therapy in Treating Patients Who Have Stage III or Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Introgen Therapeutics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: INTROGEN-201-010; CDR0000256223 (Registry Identifier: PDQ (Physician Data Query)); MDA-ID-00008
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-07

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — advexin; Docetaxel; Doxorubicin; Neoadjuvant Therapy

INTERVENTIONS:
Biological: Ad5CMV-p53 gene
Drug: docetaxel
Drug: doxorubicin hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Inserting the p53 gene into the tumor may increase the effectiveness of a chemotherapy drug by making tumor cells more sensitive to the drug. Combining chemotherapy with gene therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy with gene therapy in treating patients who have stage III or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic efficacy of docetaxel, doxorubicin, and Ad5CMV-p53 gene in patients with locally advanced breast cancer.

OUTLINE: Patients receive p53 gene by intralesional injection on days 1 and 2. Patients also receive doxorubicin IV over 15 minutes followed 1 hour later by docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 6 courses. After completion of chemotherapy, patients with a reasonable response undergo surgical resection.

PROJECTED ACCRUAL: A maximum of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage IIIA, IIIB (excluding inflammatory breast carcinoma), or IIIC OR
  * Localized stage IV
* Measurable disease
* No metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Adequate bone marrow function

Hepatic

* Adequate liver function
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Adequate kidney function

Cardiovascular

* Normal cardiac function by MUGA and/or echocardiogram

Other

* No psychological, familial, sociological, or geographical conditions that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective barrier method of contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior gene therapy using adenoviral vectors or p53 gene product

Chemotherapy

* No prior chemotherapy for breast cancer

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Van Warthood, PhD, Study Chair — Introgen Therapeutics
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States